CLINICAL TRIAL: NCT01420718
Title: Partial Pulpotomy on Caries Free Human Teeth Using iRootBP and White ProRoot MTA: a Randomized Controlled Trial
Brief Title: Partial Pulpotomy on Caries Free Human Teeth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Mahta Fazlyab, post graduate student of Endodontic department, Dental Branch, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p/439/d; IRCT201102145804N2 (Other: Iranian registry of clinical trails (IRCT))
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Dentin Bridge; Pulpitis
Keywords: partial pulpotomy; Cvek pulpotomy; MTA; iRootBP; dentin bridge
MeSH Terms: conditions — Pulpitis | interventions — Pemetrexed; iRoot BP Plus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mineral Trioxide Aggregate (Active Comparator): partial pulpotomy using White ProRoot MTA. Partial pulpotomy includes removal of 1mm of coronal pulp and covering the remaining tissue with a suitable material.
  Interventions: Drug: MTA
- iRoot BP (Experimental): Partial pulpotomy using iRoot BP. Partial pulpotomy includes removal of 1mm of coronal pulp and covering the remaining tissue with a suitable material. Bioaggregate is the first nano particle, water based root end filling material. This product includes calcium silicate, calcium hydroxide, hydroxy apatite and Tantalum oxide. Compared to MTA,this material lacks Bismuth oxide and calcium aluminate. iRoot BP is the injectable for of Bioaggregate (Injectable Root Bioaggregate Paste).
  Interventions: Drug: iRoot BP

INTERVENTIONS:
Drug: MTA — partial pulpotomy using White ProRoot MTA. Partial pulpotomy includes removal of 1mm of coronal pulp and covering the remaining tissue with a suitable material.
  Other Names: White ProRoot MTA
  Arms: Mineral Trioxide Aggregate
Drug: iRoot BP — Partial pulpotomy using iRoot BP. Partial pulpotomy includes removal of 1mm of coronal pulp and covering the remaining tissue with a suitable material. Bioaggregate is the first nano particle, water based root end filling material. This product includes calcium silicate, calcium hydroxide, hydroxy apatite and Tantalum oxide. Compared to MTA,this material lacks Bismuth oxide and calcium aluminate. iRoot BP is the injectable for of Bioaggregate (Injectable Root Bioaggregate Paste).
  Other Names: Injectable Root Bioaggregate Paste
  Arms: iRoot BP

SUMMARY:
The purpose of this study is to compare the human pulp response to partial pulpotomy using White ProRoot MTA or iRoot BP in the terms of dentinal bridge formation and inflammation.

DETAILED DESCRIPTION:
This will be a randomized single blind clinical trial. Setting and conduct: Twenty caries free premolar teeth from fifteen patients assigned for orthodontic extraction will be included. Participants including major eligibility criteria: Their parents need to sign an informed form, Patients shouldn't have any systematic complication, The teeth should be free of any symptom, caries and decalcification and should reveal a normal response to pulp sensitivity tests, No mobility or swelling in the surrounding soft tissues, sensitivity on palpation or percussion should be present. Intervention: A class one cavity will be prepared and the depth will be increased until the pulp exposure occurs. One millimeter of the coronal pulp will be removed. Then the exposure site will be covered using two pulpotomy agents: White ProRoot MTA as control group and iRoot BP. After six weeks (42 days) the teeth will be extracted after radiographic and clinical examination to find any sign of swelling, abscess or sinus tract. Main outcome measures (variables): The teeth will be sectioned and examined to compare the presence of dentinal bridge, its thickness and feature in the terms of tunnel defect formation. The underlying pulp will be assessed and graded according to the degree of inflammation as follows: grade 0 no inflammation, grade 1 mild inflammation, grade 2 moderate inflammations, grade 3 severe inflammation, grade 4 abscess formation or necrosis. Our criteria are based on ISO 7405.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are assigned to extract two premolar teeth in one jaw for orthodontic treatment plan.
* Their parents need to read and sign a fully informed form.
* They shouldn't have any systematic complication or take any medicine during the period of study.
* The teeth need to be free of any symptom, caries and decalcification
* They should give a normal response to pulp sensitivity tests (cold test) compared to the control tooth on the same quadrant.
* The teeth need to be free of mobility or swelling in the surrounding soft tissues and any sensitivity on palpation or percussion.
* On radiographic examination no apical lucency or PDL widening should be detected.

Exclusion Criteria:

* tooth crack
* tooth filling
* any caries
* hypocalcification
* The teeth showing apical lucency
* PDL widening on radiography
* sensitivity to cold, heat or bite
* The responses beyond the normal limits to pulp vitality testing
* Any medicine consumption

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
dentinal bridge formation | six weeks after intervention
  appearance of the dentinal bridge compared to normal dentin will be assessed under microscope

SECONDARY OUTCOMES:
inflammatory status of the pulp | six weeks after intervention
  microscopic evaluation : inflammatory cell count and their distribution

CONTACTS AND LOCATIONS:
Overall Officials: Mahta Fazlyab, Principal Investigator — Azad University, Dental Branch, Tehran
Locations (1):
- Azad University, Dental Branch, Tehran, Endodontic department, Tehran, Iran